CLINICAL TRIAL: NCT01434381
Title: Open Label Phase 1 Study in Malaria Naive Adults of the Safety and Immunogenicity of Pfs25-EPA/Alhydrogel, a Transmission Blocking Vaccine Against Plasmodium Falciparum
Brief Title: Initial Study of Malaria Vaccine Pfs25-EPA/Alhydrogel(Registered Trademark)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-I-N237; 11-I-N237 (Other: NIH); CIR 276 (Other: Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health)
Record Dates: First submitted 2011-09-10; First posted 2011-09-14 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Malaria
Keywords: Recombinant; Proteins; Antigen; Membrane; Assay; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pfs25-EPA/Alhydrogel (Experimental): Dose-escalation of Pfs25-EPA/Alhydrogel. Participants will receive 1 of 3 doses of Pfs25-EPA/Alhydrogel- 8 micro g, 16 micro g, or 47 micro g.
  Interventions: Biological: Pfs25-EPA/Alhydrogel

INTERVENTIONS:
Biological: Pfs25-EPA/Alhydrogel

SUMMARY:
Background:

- The malaria vaccine Pfs25-EPA/Alhydrogel may help block malaria parasites from developing in mosquitoes. When a mosquito bites a vaccinated person, the vaccine should prevent parasites from developing in the mosquito. As a result, the mosquito will not spread malaria to the next person it bites. However, the vaccine will not directly prevent people from getting sick with malaria. Researchers want to test the safety of and response to this vaccine.

Objectives:

- To test the safety of the malaria vaccine Pfs25-EPA/Alhydrogel.

Eligibility:

- Healthy volunteers between 18 and 50 years of age.

Design:

* Participants will be screened with a medical history, physical exam, and blood tests.
* They will be assigned to a study group to have either two or three doses of the vaccine. Participants will have checkups after each dose of vaccine,
* The additional doses will be given 2 months or 2 and 4 months after the first vaccine.
* Participants will have regular blood tests to check the level of the response to the vaccine.
* They will be followed for up to 1 year after the last vaccine to have any additional tests as needed.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission would be a valuable tool for local elimination or eradication of this disease. Pfs25, a surface antigen of ookinetes in the mosquito stage of P. falciparum, is a lead candidate for a malaria transmission blocking vaccine. Recombinant Pfs25 has been conjugated to Pseudomonas aeruginosa ExoProtein A (EPA), and adjuvanted with Alhydrogel(Registered Trademark). This open label, dose escalating Phase 1 study in malaria naive adults, conducted at Johns Hopkins Bloomberg School of Public Health Center for Immunization Research (CIR) in Baltimore, Maryland, will determine initial safety and immunogenicity of the vaccine given on a 2-dose,3-dose, or 4-dose schedule. Thirty (30) volunteers will be enrolled, with 5 receiving the low dose (8 micro g of conjugated Pfs25), 5 receiving the middle dose (16 micro g of conjugated Pfs25), and 20 receiving the high dose (47 micro g of conjugated Pfs25). The high dose group will receive either 2, 3 or 4 doses of vaccine, on a 0, 2, 4 and 10 month vaccination schedule. Volunteers will be followed for 12 months following the last vaccination. Safety outcomes will be local and systemic adverse events (AEs). Immunogenicity outcomes will be antibody responses as measured by ELISA, transmission blocking in a standard membrane feeding assay, and B and T cell responses.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

* Age between 18 and 50 years.
* Good general health as a result of review of medical history and/or clinical testing at the time of screening.
* Available for the duration of the trial.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* If female: subject is willing to use reliable contraception methods for the period of at least 1month (2 months for oral contraceptive pills) prior to first vaccination to 3 months after last vaccination. Reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; vaginal ring; transdermal patch; intrauterine device; abstinence; and post-menopause.

EXCLUSION CRITERIA:

A volunteer will be excluded from participating in this trial if any one of the following criteria is fulfilled:

* Pregnancy as determined by a positive urine or serum human choriogonadotropin (Beta-hCG) test at any point during the study (if female).
* Currently is lactating and breast-feeding (if female).
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
* Neutropenia as defined by an absolute neutrophil count < 1500/mm(3).
* Alanine transaminase (ALT) level above the laboratory-defined upper limit of normal.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the subject unable to comply with the protocol.
* History of receiving any investigational product within the past 30 days.
* Receipt of antimalarial prophylaxis during the past 12 months, or planned travel to a destination which would require malaria prophylaxis during the period of participation.
* Prior malaria infection by history.
* Participant has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma. This will be defined as:

  * Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years, or that requires the use of oral or parenteral corticosteroids.
  * Clinically significant reactive airway disease that does not respond to bronchodilators.
* Positive ELISA and confirmatory Western blot tests for HIV-1.
* Positive ELISA and confirmatory tests for hepatitis C virus (HCV).
* Positive hepatitis B surface antigen (HBsAg) by ELISA.
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.
* Known immunodeficiency syndrome.
* Use of chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e. prednisone > 10 mg/ day) or immunosuppressive drugs within 30 days of starting this study.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine.
* Refusal to allow storage of samples for future research.
* Any medical, psychiatric, social, or occupational condition or other responsibility that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events | All adverse events will be recorded though Day 28 after each vaccination. The frequency of systemic and local AEs will be summarized.
  Subjects will be monitored for 30 minutes following each immunization. Subjects will return to the clinic on Days 3,7,14 and 28 following each vaccination for clinical assessments, and periodically thereafter until completion

SECONDARY OUTCOMES:
To determine the antibody response to the Pfs25 protein vaccines as measured by ELISA and transmission blocking assays, and the effect on antibody responses of a third dose at four months | ELISA testing will occur on vaccination days, 2 weeks after each vaccination, and periodically until study completion

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Duffy, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Birkett AJ. PATH Malaria Vaccine Initiative (MVI): perspectives on the status of malaria vaccine development. Hum Vaccin. 2010 Jan;6(1):139-45. doi: 10.4161/hv.6.1.10462. Epub 2010 Jan 29. No abstract available. PMID 20009524
- [Background] Cheru L, Wu Y, Diouf A, Moretz SE, Muratova OV, Song G, Fay MP, Miller LH, Long CA, Miura K. The IC(50) of anti-Pfs25 antibody in membrane-feeding assay varies among species. Vaccine. 2010 Jun 17;28(27):4423-9. doi: 10.1016/j.vaccine.2010.04.036. Epub 2010 Apr 29. PMID 20434549
- [Background] Coler RN, Baldwin SL, Shaverdian N, Bertholet S, Reed SJ, Raman VS, Lu X, DeVos J, Hancock K, Katz JM, Vedvick TS, Duthie MS, Clegg CH, Van Hoeven N, Reed SG. A synthetic adjuvant to enhance and expand immune responses to influenza vaccines. PLoS One. 2010 Oct 27;5(10):e13677. doi: 10.1371/journal.pone.0013677. PMID 21060869